CLINICAL TRIAL: NCT00187226
Title: A Phase II Study of Image-Guided Radiation Therapy for Pediatric CNS Tumors and Quantification of Radiation-Related CNS Effects
Brief Title: A Study for Image-Guided Radiation Therapy in Pediatric Brain Tumors and Side Effects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT1
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Central Nervous System Tumors; Brain Tumors
Keywords: Brain neoplasm; Brain cancer; Neoplasm intracranial
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stratum 1 (Other): Ependymoma, craniopharyngioma, low-grade glioma
  Interventions: Procedure: Radiation Therapy
- Stratum 2 (Other): High-grade glioma
  Interventions: Procedure: Radiation Therapy

INTERVENTIONS:
Procedure: Radiation Therapy — External Beam Radiation Therapy: 54Gy administered at 1.8Gy per day for low-grade glioma, craniopharyngioma and selected ependymoma.
  Arms: Stratum 1
Procedure: Radiation Therapy — External Beam Radiation Therapy: 59.4Gy administered at 1.8Gy per day for high-grade glioma and selected ependymoma.
  Arms: Stratum 2

SUMMARY:
The purpose of the study was to determine if treating a limited volume of normal tissue surrounding the tumor or tumor bed using conformal radiation therapy would achieve similar rates of disease control compared to standard radiation therapy. The study was also conducted to examine the effect of irradiation on neurological, endocrine and cognitive function.

DETAILED DESCRIPTION:
Radiation therapy is commonly used to treat a variety of brain tumors in children including ependymoma, craniopharyngioma and low- and high-grade glioma. The ability of the therapy to control brain tumors in children is known to depend on the tumor type, extent of resection and other clinical factors. Children who received radiation therapy on this study were evaluated for treatment failure at 12 months. In addition to the primary objective, the study was designed to explore the association between radiation dose and volume and a variety of neurological, endocrine and cognitive deficits up to 5 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age at time of irradiation is greater than or equal to 8 months and less than or equal to 25 years
* Histologically diagnosed craniopharyngioma, ependymoma, low-grade astrocytoma or high-grade glioma and radiographically diagnosed selected patients with craniopharyngioma and low-grade glioma.
* Adequate performance status, participant has an ECOG (Performance Status Score) of 0-2(0=Normal Activity; 1=Symptoms but Ambulatory; 2=Bedridden <50% of time)
* Histologic type that requires only focal irradiation.
* No prior fractionated external beam irradiation
* Informed consent signed by patient, parent, or guardian.

Ages: 8 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 361 (Actual)
Dates: Start 1997-06 (Actual); Primary Completion 2005-03-31 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Merchant, D.O., Ph.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Netson KL, Conklin HM, Wu S, Xiong X, Merchant TE. Longitudinal investigation of adaptive functioning following conformal irradiation for pediatric craniopharyngioma and low-grade glioma. Int J Radiat Oncol Biol Phys. 2013 Apr 1;85(5):1301-6. doi: 10.1016/j.ijrobp.2012.10.031. Epub 2012 Dec 11. PMID 23245284
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 202 patients were enrolled between July 11, 1997 and January 14, 2003 for the therapeutic phase of the trial. Among those patients, 167 were treated with a 1cm clinical target volume (CTV) margin and 35 were treated with a 2cm CTV margin. Local tumor progression was determined by MR imaging.
  202 patients correspond to the initial number of patients enrolled prior to the amendment which increased accrual 361
Groups:
- 1cm Clinical Target Volume Margin - Ependymoma: Patients with Ependymoma in the 1cm clinical target volume margin group.
- 1cm Clinical Target Volume Margin - Low-grade Glioma: Patients with Low-grade Glioma in the 1cm clinical target volume margin group.
- 1cm Clinical Target Volume Margin - Craniopharyngioma: Patients with Craniopharyngioma in the 1cm clinical target volume margin group.
- 1cm Clinical Target Volume Margin - Other: Remaining patients in the 1cm clinical target volume margin group.
- 2cm Clinical Target Volume Margin - High-grade Glioma: Patients with High-grade glioma in the 2cm clinical target volume margin group.
- 2cm Clinical Target Volume Margin - Low-grade Glioma: Patients with Low-grade Glioma in the 2cm clinical target volume margin group.
Period: Overall Study
Arm/Group | 1cm Clinical Target Volume Margin - Ependymoma | 1cm Clinical Target Volume Margin - Low-grade Glioma | 1cm Clinical Target Volume Margin - Craniopharyngioma | 1cm Clinical Target Volume Margin - Other | 2cm Clinical Target Volume Margin - High-grade Glioma | 2cm Clinical Target Volume Margin - Low-grade Glioma
Started | 88 | 49 | 28 | 2 | 34 | 1
Completed | 88 | 49 | 28 | 2 | 34 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1cm Clinical Target Volume Margin - Ependymoma | 1cm Clinical Target Volume Margin - Low-grade Glioma | 1cm Clinical Target Volume Margin - Craniopharyngioma | 1cm Clinical Target Volume Margin - Other | 2cm Clinical Target Volume Margin - High-grade Glioma | 2cm Clinical Target Volume Margin - Low-grade Glioma | Total
Number analyzed (Participants) | 88 | 49 | 28 | 2 | 34 | 1 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86 | 48 | 28 | 2 | 26 | 1 | 191
  Between 18 and 65 years | 2 | 1 | 0 | 0 | 8 | 0 | 11
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 24 | 16 | 1 | 16 | 0 | 98
  Male | 47 | 25 | 12 | 1 | 18 | 1 | 104

OUTCOME MEASURES:

1. Primary Outcome: Local Tumor Control
Description: Local tumor control was determined by Magnetic Resonance Imaging (MRI) of the brain and spine performed after radiation therapy. Imaging studies were performed every 3-4 months during the first three years and then every 6 months through five years. Imaging studies demonstrating tumor progression were electronically registered to the imaging data used to plan therapy. Local failure included tumor progression within the volume that received the prescribed dose of irradiation.
Time Frame: 12 months after the enrollment of the last therapeutic patient
Population: Patients with Ependymoma, Craniopharyngioma, Low-grade Glioma, and High-grade Glioma were analyzed by diagnosis.
Measure: Log Mean (95% Confidence Interval); unit: Proportion of patients
Arm/Group | 1cm Clinical Target Volume Margin - Ependymoma | 1cm Clinical Target Volume Margin - Low-grade Glioma | 1cm Clinical Target Volume Margin - Craniopharyngioma | 1cm Clinical Target Volume Margin - Other | 2cm Clinical Target Volume Margin - High-grade Glioma | 2cm Clinical Target Volume Margin - Low-grade Glioma
Number analyzed (Participants) | 88 | 49 | 28 | 2 | 34 | 1
Proportion of patients | 0.966 [0.904 to 0.993] | 0.959 [0.860 to 0.995] | 1.000 [0.877 to 1.000] | 1.000 [1.000 to 1.000] | 0.618 [0.436 to 0.778] | 1.000 [1.000 to 1.000]

ADVERSE EVENTS:
Time Frame: Patients enrolled on this study included 202 patients who were enrolled between July 11, 1997 and January 14, 2003. Patients are followed 30 days post off-study.
Arm/Group | 1cm Clinical Target Volume Margin - Ependymoma | 1cm Clinical Target Volume Margin - Low-grade Glioma | 1cm Clinical Target Volume Margin - Craniopharyngioma | 1cm Clinical Target Volume Margin - Other | 2cm Clinical Target Volume Margin - High-grade Glioma | 2cm Clinical Target Volume Margin - Low-grade Glioma
Serious Adverse Events (participants affected / at risk) | 1/88 | 0/49 | 2/28 | 0/2 | 1/34 | 0/1
Other Adverse Events (participants affected / at risk) | 9/88 | 4/49 | 0/28 | 0/2 | 0/34 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1cm Clinical Target Volume Margin - Ependymoma (N=88) | 1cm Clinical Target Volume Margin - Low-grade Glioma (N=49) | 1cm Clinical Target Volume Margin - Craniopharyngioma (N=28) | 1cm Clinical Target Volume Margin - Other (N=2) | 2cm Clinical Target Volume Margin - High-grade Glioma (N=34) | 2cm Clinical Target Volume Margin - Low-grade Glioma (N=1)
CNS Ischemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1cm Clinical Target Volume Margin - Ependymoma (N=88) | 1cm Clinical Target Volume Margin - Low-grade Glioma (N=49) | 1cm Clinical Target Volume Margin - Craniopharyngioma (N=28) | 1cm Clinical Target Volume Margin - Other (N=2) | 2cm Clinical Target Volume Margin - High-grade Glioma (N=34) | 2cm Clinical Target Volume Margin - Low-grade Glioma (N=1)
Infection (Infections and infestations) | 9 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuromotor (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes